CLINICAL TRIAL: NCT04293419
Title: Phase II Study of Durvalumab (MEDI4736) Plus Total Neoadjuvant Therapy (TNT) in Locally Advanced Rectal Cancer (The DUREC Trial)
Brief Title: Durvalumab (MEDI4736) Plus Total Neoadjuvant Therapy (TNT) in Locally Advanced Rectal Cancer
Acronym: DUREC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Grupo Espanol Multidisciplinario del Cancer Digestivo (Other)
Collaborators: AstraZeneca (Industry); Vall d'Hebron Institute of Oncology (VHIO) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESR-17-13082
Record Dates: First submitted 2020-02-13; First posted 2020-03-03 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — durvalumab

STUDY DESIGN:
Intervention Model Description: Patients will be included following inclusion/exclusion criteria in a prospective, non-randomized, open label, single arm phase II study to receive 6 cycles of mFOLFOX6 (oxaliplatin, leucovorin and fluorouracil) followed by long course chemoradiotherapy (50.4 Gy together with capecitabine) followed by surgery. Patients will receive durvalumab 1500 mg every 4 weeks during induction chemotherapy, chemoradiotherapy and waiting period until surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Durvalumab (MEDI4736) — 6 cycles of mFOLFOX6 (oxaliplatin, leucovorin and fluorouracil) followed by long course chemoradiotherapy (50.4 Gy together with capecitabine) followed by surgery. Patients will receive durvalumab 1500 mg every 4 weeks during induction chemotherapy, chemoradiotherapy and waiting period until surgery.

SUMMARY:
The addition of durvalumab to total neoadjuvant therapy (TNT) in locally advanced rectal cancer may improve the pathological complete response rate. The induction platinum-based chemotherapy may increase the neoantigen formation together with the chemoradiotherapy period. Starting durvalumab during the first chemotherapy session and continuing during the 6-week period of chemoradiotherapy could change and create the needed environment to increase the efficacy of durvalumab in this setting. Additionally, the 8-12 week rest period from the end of the chemoradiotherapy and the radical surgery, treatment with durvalumab may continue improving the response and outcome of patients without jeopardizing the surgery (which needs this period out of chemotherapy and radiotherapy to avoid postoperative complications, but not for anti-PDL-1 therapy).

Patients will be included following inclusion/exclusion criteria in a prospective, non-randomized, open label, single arm phase II study to receive 6 cycles of mFOLFOX6 (oxaliplatin, leucovorin and fluorouracil) followed by long course chemoradiotherapy (50.4 Gy together with capecitabine) followed by surgery. Patients will receive durvalumab 1500 mg every 4 weeks during induction chemotherapy, chemoradiotherapy and waiting period until surgery.

DETAILED DESCRIPTION:
The DUREC trial comprises three treatment periods: induction chemotherapy, chemoradiotherapy and waiting period until surgery.

Durvalumab (MEDI4736) will be supplied in glass vials containing 500 mg of liquid solution at a concentration of 50 mg/mL for intravenous(IV) administration. Flat dose of 1500 mg every 4 weeks will be administered during induction chemotherapy, chemoradiotherapy and waiting period until surgery.

Induction chemotherapy (Week 1-12) Patients will be treated with Durvalumab and FOLFOX6 regimen. Modified FOLFOX6 regimen consists of 2-hour infusion of oxaliplatin (85 mg/m2) and 2-hour infusion of leucovorin (400 mg/m2) on Day l, followed by 5-fluorouracil (5-FU) bolus (400 mg/m2) on Day 1 and 44-hour on continuous infusion (2400 mg/m2). FOLFOX6 regimen will be repeated at 2-week intervals.

Chemoradiotherapy (Week 13-20) Patients will be treated with Durvalumab, radiotherapy and capecitabine. All patients will receive 28 daily (5/7 days) fractions of 1.8 Gy up to a total dose of 50.4 Gy to the pelvic field including the tumour bed with a margin and the regional lymph nodes.

Capecitabine will be given during radiotherapy in a dose of 825 mg/m2 bid (twice per day) 7/7 days during all radiotherapy period (38 days approximately, considering bank holidays and radiotherapy machinery periodic revisions) Waiting period until surgery (21-31) Patients will be treated with Durvalumab on week 21 and 25. To assess the tolerability and toxicity profile of the combination of mFOLFOX6 + durvalumab and CRT + durvalumab the investigators plan to perform a run-in treatment phase including the first 6 patients in the study and stop recruitment until the last of these 6 patients will be operated and 30-days postsurgery period will be completed. If 2 or less dose limiting toxicities (DLTs) related with durvalumab therapy are observed in these 6 patients, recruitment will be opened again to reach the planned 58 patients.

ELIGIBILITY:
Inclusion Criteria:

- 1) Written informed consent obtained from the patient prior to performing any protocol-related procedures, including screening evaluations.

2) Age > 18 years at time of study entry. 3) Must have a life expectancy of at least 12 weeks 4) Eastern Cooperative Oncology Group (ECOG)performance status of 0 or 1. 5) Body weight >30kg. 6) Biopsy-proven, newly diagnosed primary rectal adenocarcinoma, with the lowest part of the tumour less than 12 cm from the anal verge using a rigid rectoscope or flexible endoscope.

7) Mandatory tumour and blood samples for translational research. 8) High risk MRI-defined rectal cancer: Presence of at least 1 of the following on high resolution, thin-slice MRI (3 mm): Upper-Middle Third Tumours

-mrT3

1. Extramural vascular invasion (EMVI) positive
2. Extramural extension > 5 mms into perirectal fat
3. Mesorectal fascia (MRF) threatened or involved (tumour or lymph node < 1mm from MRF) -mrT4 Distal Third Tumours (≤5 cm from anal verge) - mrT3 tumour at or below levators - T4 as above N2(≥4 lymph nodes at mesorectum radiologically suggestive of metastatic lymph nodes) 9) No contraindications to chemotherapy and radiotherapy 10) Adequate normal organ and marrow function as defined below:

   - Haemoglobin ≥9.0 g/dL.

   - Absolute neutrophil count (ANC) >1500 per mm3.

   - Platelet count ≥100,000 per mm3.
   * Serum bilirubin ≤1.5 x institutional upper limit of normal (ULN). This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician.
   * AST (SGOT)/ALT (SGPT) ≤2.5 x institutional upper limit of normal.
   * Measured creatinine clearance (CL) >40 mL/min or Calculated creatinine CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance:

   Males:

   Creatinine CL (mL/min) = Weight (kg) x (140 - Age) 72 x serum creatinine (mg/dL)

   Females:

   Creatinine CL (mL/min) = Weight (kg) x (140 - Age) x 0.85 72 x serum creatinine (mg/dL) 11) Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

   - Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
   * Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).

     12) Patients willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

   Exclusion Criteria:
   * 1) Participation in another clinical study with an investigational product during the last 6 months.

     2) Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study.

     3) Prior therapy for rectal cancer. 4) Presence of metastatic disease or recurrent rectal tumour. Familial Adenomatosis Polyposis coli (FAP), Hereditary Non-Polyposis Colorectal Cancer (HNPCC), active Crohn's disease or active ulcerative Colitis.

     5) Extensive growth into cranial part of the sacrum (above S3) or the lumbosacral nerve roots indicating that surgery will never be possible even if substantial tumour down-sizing is seen.

     6) Known DPD deficiency. 7) Persistent peripheral neural toxicity > grade 2. 8) Intestinal occlusion. Patients with intestinal occlusion due to the primary rectal tumour, that could participate in the study, may be included after a derivative intestinal surgery.

     9) Any previous treatment with a PD1 or PD-L1 inhibitor, including durvalumab. 10) Mean QT interval corrected for heart rate (QTc) ≥470 ms calculated from 3 electrocardiograms (ECGs) using Fridericia's Correction.

     11) Current or prior use of immunosuppressive medication within 28 days before the first dose of durvalumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid. The following are exceptions to this criterion:
   * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection).
   * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent.
   * Steroids as premedication for hypersensitivity reactions (e.g.,CT scan premedication).

     12) Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria
   * Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician.
   * Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with the Study Physician.

     13) Any concurrent chemotherapy, IP, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.

     14) Previous radiotherapy in the pelvic region (e.g. prostate) or previous rectal surgery (e.g.TEM).

     15) History of allogenic organ transplantation. 16) Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:
   * Patients with vitiligo or alopecia
   * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
   * Any chronic skin condition that does not require systemic therapy
   * Patients without active disease in the last 5 years may be included but only after consultation with the study physician
   * Patients with celiac disease controlled by diet alone 17) Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent 18) History of another primary malignancy except for
   * Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of IP and of low potential risk for recurrence
   * Adequately treated non-melanoma skin cancer or lentigomaligna without evidence of disease
   * Adequately treated carcinoma in situ without evidence of disease 19) History of active primary immunodeficiency 20) Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.

     21) Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note: Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 30 days after the last dose of IP.

     22) Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 180 days after the last dose of durvalumab monotherapy.

     23) Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.

     24) Judgment by the investigator that the patient is unsuitable to participate in the study and the patient is unlikely to comply with study procedures, restrictions and requirements.

     25) Known allergy or hypersensitivity to IP or any excipient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2019-12-18 (Actual); Primary Completion 2024-12-18 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) rate | Immediately after the surgery

SECONDARY OUTCOMES:
Tumor downstaging | Will be assessed during the 3-year period of follow-up
Tumor regression grade (TRG) | Will be assessed during the 3-year period of follow-up
R0 resection rate | Immediately after the surgery
Clear circumferential resection margin (CRM) rate | Immediately after the surgery
3-year disease-free survival (DFS) | 3 years after the surgery
Toxicity profile (short and long term) | From date of randomization until three years after surgery, assessed up to 44 months
Surgical complications | Immediately after the surgery
Calculation of the neoadjuvant rectal (NAR) score | Immediately after the surgery

CONTACTS AND LOCATIONS:
Locations (10):
- Spain (10):
  - Parc Taulí, Sabadell, Barcelona
  - H. Moises Broggi, Sant Joan Despí, Barcelona
  - H. Navarra, Pamplona, Navarre
  - Complejo Hospitalario Universitario A Coruña (CHUAC), A Coruña
  - Hospital Vall d'Hebron, Barcelona
  - H. Clínic Barcelona, Barcelona
  - H. de Elche, Elche
  - H. 12 de Octubre, Madrid
  - Instituto Valenciano de Oncología (IVO), Valencia
  - H. Miguel Servet Zaragoza, Zaragoza

IPD SHARING:
Plan to Share IPD: No